CLINICAL TRIAL: NCT04563728
Title: Leveraging Surveillance Technology to Improve Safety in Community Aging Populations
Brief Title: Use Surveillance Technology to Reduce Elder Abuse Recidivism
Acronym: MC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Rutgers University (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro2019001409
Record Dates: First submitted 2020-03-30; First posted 2020-09-24 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Elder Abuse; Self Neglect; Aging; Domestic Abuse

STUDY DESIGN:
Intervention Model Description: Three groups of people receive different interventions and usual care.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Comparing two different intervention strategies, participants and research assistants will be masked about the assignment during the 8-week participation. In the camera and mock camera group, participants will not be told which group they are a part of. In either the camera or mock camera group, research assistants (RAs) administering consent will also not be told which group the participant is a part of to avoid accidental reveal of groups. Groups will be revealed at the end of the study participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Camera Group (Active Comparator): 1) The camera(s) will be a stationary device installed by the study technician on the ceiling of a common living area of the participant's home. The camera(s) will record video and audio data to be stored in our secure data base. The cameras will be purchased from YI Technology (see more details in Section 1.7). A sign will be placed outside the home to notify individuals regarding the potential recording, reading, "NOTICE Audio and/or video surveillance may be in use on these premises". Highlighted video and audio data will be reviewed daily by the study technician. If there is evidence of abuse, exploitation, and neglect on these video and audio data, a report will be made to APS and the IRB.
  Interventions: Behavioral: Surveillance camera(s)
- Mock Camera Group (Active Comparator): 2) The mock camera(s) will be a stationary device installed on the ceiling of a common living area of the participant's home. They will not record video or audio but will be installed with a sensor chip and a Wi-Fi connection, which will notify the study team if the device has been touched, tampered, altered, or disrupted power sources. After installing the device, the study technician and study coordinator will test the anti-tampering sensor to ensure potential future tampering will be detected. A sign will be placed outside the home to notify individuals regarding the potential recording, reading, "NOTICE Audio and/or video surveillance may be in use on these premises". Daily check-ins to assess whether elder abuse may have been experienced by the participant will occur by phone or other preferred mode of communication. In the event of reported abuse, exploitation, and neglect, despite not being mandatory reporters, we will report to NJ APS and the IRB.
  Interventions: Behavioral: Surveillance camera(s)
- Usual Care (No Intervention): Each participant will receive educational packages about elderly community-living.

INTERVENTIONS:
Behavioral: Surveillance camera(s) — the mock camera intervention is for testing whether the impression of surveillance would have the effect to reduce the recidivism of elder abuse in home settings; 2) whether less costly options (mock cameras) are as effective as surveillance camera(s) in reducing the recidivism of elder abuse; 3) feasibility and acceptability of surveillance camera(s)
  Arms: Camera Group; Mock Camera Group

SUMMARY:
The project is to build multi-sector and multi-institutional partnerships to test the feasibility, acceptability, and efficacy of a pilot surveillance camera intervention (N=10) to reduce the frequency and severity of abuse, exploitation, and neglect in community older adults.

DETAILED DESCRIPTION:
This a feasibility investigation that aims to conduct an 8-week pilot RCT (N=10 total) to test the potential effectiveness of a surveillance intervention to reduce frequency and severity of elder abuse among older populations. Eligible participants will be recruited from community-dwelling populations in which an older adult victim has experienced elder abuse (abuse, exploitation, neglect) according to New Jersey APS referrals or our screening. With informed written consent, participants will be evenly randomized into one of three conditions: camera, mock camera, and control (usual care).

Primary outcomes are elder abuse cases including psychological, physical, sexual abuse, financial exploitations, caregiver neglect, and self-neglect measured by 83 items. For psychological and physical abuse, we use eight items and ten items from a modified Conflict Tactics Scale (CTS).46-53. Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice.54 Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living among individuals living with at least one person.35,55 Self-neglect was assessed by a widely used and validated measurement56,57.The measurement was reviewed by a community advisory board of over 20 community organizations led by a geriatrician and has shown good contend, convergent58, and predictive validity59.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 or older;
2. Community-living;
3. Individuals identified by New Jersey APS as potentially at risk of elder abuse; OR Individuals who have experienced abuse, exploitation, or neglect within the last 3 months (assessed by any "present" or "yes" response to elder abuse questions on the screener).

Exclusion Criteria:

1. Live in institutional and/or residential facilities;
2. Have plans to move for the next 3 months;
3. Unable to understand and provide written consent. Capacity to consent will be determined by a score of at least 24 on the Mini-mental state examination;
4. Have impairment in eating, dressing, bathing, walking, transferring, grooming, bladder control, or toileting. These will be determined by any "present" or "positive" item on the Activities of Daily Living (ADLs).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
elder abuse prevalence | Baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | First week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Second week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Third week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Fourth week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Fifth week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Sixth week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Seventh week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Eighth week of participation
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Tenth week since baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Third month since baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Fourth month since baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Fifth month since baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.
elder abuse incidence | Sixth month since baseline
  Psychological, physical, sexual abuse, financial exploitation, caregiver neglect, and self-neglect. For psychological and physical abuse, we will use 8 items and 10 items from a modified Conflict Tactics Scale (CTS). Sexual abuse will be assessed by a question asking about experiences of being touched in private areas when unwanted. Financial exploitation will be assessed by the 17-item Financial Exploitation Scale, adapted from Conrad et al in a study funded by the Department of Justice. Caregiver neglect will be assessed by 20 items of unmet needs in key activities of daily living. Self-neglect will be assessed by a validated 25-item measurement.
  Items will be combined to report whether any vs no abuse/neglect/exploitation was experienced. In addition, multiple definitions of severity can be determined by combining these instruments and using various cut off points to determine severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Institute for Health, Health Care Policy and Aging Research, New Brunswick, New Jersey, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT04563728/ICF_000.pdf